CLINICAL TRIAL: NCT06704516
Title: COmmencing Menopausal HOrmone Replacement Therapy and the Effect on Metabolic-dysfunction Associated Steatotic Liver Disease: a Pilot Mechanistic Study
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: Oxford University Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 345429
Record Dates: First submitted 2024-10-29; First posted 2024-11-26 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Menopause; Metabolic Dysfunction Associated Steatotic Liver Disease
Keywords: hormone; MASLD; NAFLD; liver; estrogen; replacement; adipose; oestrogen; fat; MASH; steatosis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Platelet Glycoprotein IV Deficiency; Fatty Liver | interventions — Hormone Replacement Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Hormone Replacement Therapy (Experimental): Participants starting any brand, composition, route and dose of oestrogen-based systemic hormone replacement therapy, will be included in this group.
  Interventions: Drug: Menopausal hormone therapy

INTERVENTIONS:
Drug: Menopausal hormone therapy — Any brand, composition, route and dose of systemic menopausal hormone therapy containing oestrogen.
  Brands of HRT include oestrogel, Evorel, Lenzetto, Estradot, Progynova (this list is not exhaustive)

SUMMARY:
Metabolic dysfunction-associated steatotic liver disease (MASLD) is the most common cause of chronic liver disease worldwide, currently affecting approximately 1-in-4 people globally. The prevalence is expected to rise further, driven at least partly by the epidemic of obesity and diabetes. MASLD is a condition of fat build-up in the liver that can progress to liver scarring which is associated with higher chances of death. Women are more than twice as likely to develop MASLD after menopause compared to before menopause, and previous research has shown that this may be caused by a lack of oestrogen. A lack of oestrogen is also believed to lead to harmful changes in adipose (body fat), which has an important role in the development of MASLD. Oestrogen contained in hormone replacement therapy (HRT) is an effective treatment for hot flushes and other problems in menopause. The popularity of HRT has increased dramatically in the United Kingdom in recent years, however the exact way in which it affects adipose and MASLD is unclear. The investigators will study how HRT affects the processes that drive MASLD in 10 women before and after using the treatment. This is a small-scale pilot study to understand feasibility of recruitment and test the procedures for a future, larger-scale studies.

The investigators will recruit women who are about to begin HRT for the first time and perform the same tests for each participant before starting HRT, and after using HRT for 12-weeks. The participants will undergo meal testing including non-radioactive, stable isotopes, and blood and breath samples will be collected to measure fat processing. The total fat content of the liver will be measured using magnetic resonance imaging (MRI) scans. Adipose samples will be collected, fat metabolites will be measured and the distribution of fat around the body will be assessed using a dual energy x-ray absorptiometry (DEXA) scan. To find out how HRT affects these processes, the results from before and after using HRT will be compared. Understanding how HRT affects adipose and the liver may help reduce the development of MASLD in women after the menopause and improve their health and survival.

ELIGIBILITY:
Inclusion Criteria:

* Potential participant is willing and able to give informed consent for participation in the trial
* In the Investigator's opinion, is able and willing to comply with all trial requirements
* Female, aged 18 years and above
* Body mass index 18 to 45 kg/m2
* Postmenopausal status:

  * For women ≥ 40 defined clinically (amenorrhoea for ≥ 1 year) or biochemically (FSH >30IU/L on 2 occasions 4-6 weeks apart).
  * For women < 40 defined as a combination of oligomenorrhoea/amenorrhoea for ≥ 4 months and FSH >30IU/L on 2 occasions 4-6 weeks apart
  * Women who have undergone bilateral oophorectomy (no additional testing is required)
* Low oestradiol levels
* No exposure to systemic oestrogen-based HRT within the previous 3 months
* Willing to allow his or her General Practitioner and consultant, if appropriate, to be notified of participation in the trial.

Exclusion Criteria:

* Potential participant with known chronic liver disease, with the exception of MASLD
* The use of drugs which, in the opinion of the investigator, will significantly impact on hepatic lipid content or metabolism. This applies to drugs currently being used or used in the past, within a timeframe where the investigator believes it may impact hepatic lipid content or metabolism.
* Potential participant with any other medical explanation for amenorrhoea, apart from menopause
* History of harmful alcohol consumption (>35 units/week) or alcohol misuse disorder
* Potential participants with contraindication to MRI
* Scheduled elective surgery or other procedures requiring general anaesthesia during the trial.
* Any other significant disease or disorder which, in the opinion of the Investigator, may either put the participants at risk because of participation in the trial, or may influence the result of the trial, or the participant's ability to participate in the trial.
* Potential participant with life expectancy of less than 6 months.
* Potential participants who have participated in another research trial involving an investigational product in the past 12 weeks.
* Potential participants without a sufficient understanding of written or verbal English to participate in the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2025-08-05 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Recruitment into an experimental medicine study investigating the impact of HRT on MASLD | 7 months
  Number of participants who are screened and recruited into the study

SECONDARY OUTCOMES:
Acceptability of experimental protocols in experimental medicine study investigating the impact of HRT on MASLD | From enrollment to the end of the study after completing 12 weeks of intervention
  Feedback from questionnaire completed by study participants
Participant retention in an experimental medicine study investigating the impact of HRT on MASLD | From enrollment to the end of the study after completing 12 weeks of intervention
  Number of participants who complete the study (per protocol)
Fatty acid esterification into triglyceride | Performed at baseline and after 12 weeks of intervention
  Measurement of 13C-palmitate incorporation into very low density lipoprotein triglyceride (VLDL-TG)
Hepatic lipid content | At baseline and after 12 weeks of intervention
  Measurement of intrahepatic triglyceride content by magnetic resonance imaging / spectroscopy
Whole body fatty acid oxidation | At baseline and after 12 weeks of intervention
  Measurement of incorporation of 13C into breath CO2 using GC-C-IRMS.
Fasting and postprandial plasma intrahepatic fatty acid synthesis. | At baseline and after 12 weeks of intervention
  Change in hepatic fatty acid synthesis as measured by incorporation of 2H2 palmitate (via 2H2O) into VLDL-TG
Liver profile blood tests and circulating lipid profiles | At baseline and after 12 weeks of intervention
  Routine laboratory biochemistry
Interstitial levels of metabolites in adipose tissue | At baseline and after 12 weeks of intervention
  Change in adipose tissue metabolite profile
Adipose tissue transcriptomic profile | At baseline and after 12 weeks of intervention
  Change in adipose tissue transcriptomic profile in abdominal subcutaneous and gluteal depots
Total and regional lean and fat tissue distribution | At baseline and after 12 weeks of intervention
  Total and regional lean and fat mass on Dual energy X-ray absorptiometry (DXA) scan

OTHER OUTCOMES:
Adipose tissue steroid profile | At baseline and after 12 weeks of intervention
  Adipose tissue steroid profile

CONTACTS AND LOCATIONS:
Locations (1):
- Oxford Centre for Diabetes Endocrinology and Metabolism (OCDEM), Churchill Hospital, Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No